CLINICAL TRIAL: NCT04611698
Title: Immediate Loading of Bone Anchored Hearing Devices
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Manchester University NHS Foundation Trust (Other Government)
Collaborators: Northern Care Alliance NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: R03963
Record Dates: First submitted 2020-10-22; First posted 2020-11-02 (Actual); Last update posted 2023-04-25 (Actual); Status verified 2023-04

CONDITIONS: Hearing Loss
MeSH Terms: conditions — Hearing Loss

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immediate loading group (Experimental): Visit 1 Implant surgery + Device loading Baseline Visit 2 Followup examination 2 weeks (2/+ 5 days) Visit 3 Followup examination 3 months (± 1 week) Visit 4 Followup examination 6 months (± 1 week) Visit 5 Followup examination 12 months (± 1 month)
  Interventions: Device: Baha sound processor BA400
- 2-week loading group (Experimental): Visit 1 Implant surgery Baseline Visit 2 Device loading 2 weeks (2/+5 days) Visit 3 Followup examination 3 months (± 1 week) Visit 4 Followup examination 6 months (± 1 week) Visit 5 Followup examination 12 months (± 1 month)
  Interventions: Device: Baha sound processor BA400

INTERVENTIONS:
Device: Baha sound processor BA400 — Baha sound processor BA400 is a cochlear implant designed specifically for soft tissue preservation.

SUMMARY:
Bone anchored hearing aids provide a hearing solution for patients that are unable to wear traditional air conduction hearing aid solutions. The technology of the devices has developed significantly over the last 510 years and patients are gaining access to their sound processor at a much earlier stage than when first brought onto the market. Despite this the investigators feel there is still room to develop this and with the new abutments with specialised hydroxyapatite coating it is hoped that patients can be loaded with their sound processor in the day of surgery. This study will compare abutment stability between two groups of patients. Those loaded immediately with their sound processor and those loaded traditionally at 2 weeks post operatively.

At routine followup appointments patients will have the stability of their abutment checked and the investigators will compare to see if loading earlier had any detrimental effects on osteointegration and the stability of the abutment.

Based on the favourable outcomes and high stability record for the BA400 it is anticipated that the time to processor fitting may be further reduced, provided favourable bone conditions at the implant site and provided satisfactory soft tissue status at the time of loading. It is hypothesised that loading immediately at the time of surgery is possible with comparable short and long term outcomes when compared to standard loading at 2 weeks

ELIGIBILITY:
Inclusion Criteria:

* Patients eligible for receiving the Baha system.

Exclusion Criteria:

* Adult patients, i.e. ≥18 years
* Eligible for the Baha system
* Bone thickness at the implant site of at least 4 mm
* No known disease or treatment that compromises / will compromise the bone quality at the implant site

Ages: 18 Years to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
Compare device stability and rate of successful implantation | 12 months
  Measuring device stability and rate of successful implantation for patients fitted with the Baha BA400 immediately on the day of surgery and at fitting 2 weeks post operatively. A successful implant is an implant that osseointegrates and is stable over time when supporting the load of the Baha sound processor.

SECONDARY OUTCOMES:
Measure the stability, as determined by Implant Stability Quotient (ISQ) values, of Baha implants placed immediately and at 23 weeks post operatively. | 23 weeks
Record implant survival over time. | 12 months
Monitor the status of the periimplant soft tissue using the classification proposed by Holgers' et al. | 12 months

IPD SHARING:
Plan to Share IPD: No